CLINICAL TRIAL: NCT04448964
Title: A Randomized, Open-Label, 3-way Cross-over (Part 1) and 2-way Cross-over (Part 2) Study in Healthy Participants to Evaluate the Relative Bioavailability and the Food Effect of an Oral Tablet Formulation Relative to a Capsule Formulation of JNJ-70033093
Brief Title: A Study of JNJ-70033093 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108803; 2020-000565-17 (EudraCT Number); 70033093THR1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-06-25; First posted 2020-06-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part 1: Treatment Sequence ABC (Experimental): Participants will receive a single dose of JNJ-70033093 spray-dried dispersion (SDD) tablet under fasted conditions (Treatment A) in Treatment Period 1, followed by JNJ-70033093 SDD tablet in fed conditions (Treatment B) in Treatment Period 2, and then JNJ-70033093 SDD granule capsule under fasted conditions (Treatment C) in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 1: Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment C in Treatment Period 2, and then Treatment A in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 1: Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment A in Treatment Period 2, and then Treatment B in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 1: Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1, followed by Treatment C in Treatment Period 2, and then Treatment B in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 1: Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2, and then Treatment C in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 1: Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2, and then Treatment A in Treatment Period 3 on Day 1 of each Period during Part 1. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence DE (Experimental): Participants will receive Treatment D (single dose of JNJ-70033093 SDD tablet in fed conditions) in Treatment Period 1, and then Treatment E (single dose of JNJ-70033093 SDD granule capsule under fasted conditions) in Treatment Period 2 on Day 1 of each Period during Part 2. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093
- Part 2: Treatment Sequence ED (Experimental): Participants will receive Treatment E in Treatment Period 1, and then Treatment D in Treatment Period 2 on Day 1 of each Period during Part 2. There will be a wash-out period of at least 5 days and up to 2 weeks between Day 1 of each treatment period.
  Interventions: Drug: JNJ-70033093

INTERVENTIONS:
Drug: JNJ-70033093 — JNJ-70033093 will be administered orally as per assigned treatment sequence.
  Other Names: BMS-986177

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and relative bioavailability of a single dose of JNJ-70033093 spray dried dispersion (SDD) tablets compared with JNJ-70033093 SDD granule capsules in healthy participants under fasting conditions in Part 1 and 2 and to assess the effect of food on the bioavailability of a single dose of JNJ-70033093 SDD tablets in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and on Day -1 of Treatment Period 1. If there are abnormalities, the investigator may decide that the abnormalities or deviations from normal are not clinically significant, in which case the participant may be included
* Healthy on the basis of safety laboratory tests performed at screening and on Day -1 of Period 1. If the results of the safety laboratory tests are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant
* If a woman, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and urine pregnancy test on Day 1 of each treatment period
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2), and body weight not less than 50 kg at screening
* After being supine for 5 minutes, systolic blood pressure between 90 and 140 millimeter of Mercury (mmHg), inclusive; and no higher than 90 mmHg diastolic blood pressure at screening and on Day -1 of Treatment Period 1
* Must sign an ICF indicating that they understand the purpose of, and procedures required for the study and is willing to participate in the study
* Before randomization, a woman must be either: a.) Not of childbearing potential (Postmenopausal- no menses for 12 months without an alternative medical cause and Permanently sterile- include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy); b.) of childbearing potential and practicing a highly effective method of contraception for at least 3 months prior to the study entry and agrees to remain on a highly effective method of contraception throughout the study and for at least 34 days after the last dose of study drug
* During the study, a man who is sexually active with a woman of childbearing potential or with a woman who is pregnant must agree to use a barrier method of contraception

Exclusion Criteria:

* History of any known illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments.
* History of any clinically significant drug or food allergies (such as anaphylaxis or hepatotoxicity) and known allergy to the study drugs or any of the excipients of the formulation
* History of allergy to or unwillingness to consume any component of the standardized high-fat breakfast menu to be provided in this study
* Use of any systemic strong cytochrome P450 P glycoprotein ([CYP] 3A4/P-gp) inducers (example, [rifampin]) or inhibitors (example, [itraconazole]) within 4 weeks before the first dose of the study drug
* Participants with current hepatitis B infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C infection (confirmed by hepatitis C virus [HCV] antibody), or human immunodeficiency virus type 1 (HIV-1) or human immunodeficiency virus type 2 (HIV-2) infection at study screening
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry or urinalysis at screening or on Day -1 of Treatment Period 1 as determined by the investigator or appropriate designee
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for hormonal contraceptives, hormone replacement therapy and paracetamol (acetaminophen) within 14 days before the first dose of the study drug until completion of the study
* Any of the following on a 12-lead electrocardiogram (ECG) and the assessment of QT interval, confirmed by repeat at screening and Day -1 of Treatment Period 1: a.) Heart rate greater than (>) 100 beats per minute (bpm); b.) PR > 210 milliseconds (ms); c.) QRS > 120 ms; d.) QT corrected according to Fridericia's formula (QTcF) > 450 ms for male and > 470 ms for female

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-70033093 | Up to 72 hours post dose
  Cmax is defined as maximum observed plasma concentration after administration of JNJ-70033093.
Part 1 and 2: Area Under the Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC [0-last]) of JNJ-70033093 | Up to 72 hours post dose
  AUC (0-last) is defined as area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration after administration of JNJ-70033093.
Part 1 and 2: Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC [0-inf]) of JNJ-70033093 | Up to 72 hours post dose
  AUC (0-inf) is defined as area under the plasma concentration-time curve from time 0 to infinity after administration of JNJ-70033093.
Part 1 and 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-70033093 | Up to 72 hours post dose
  Tmax is defined time to reach the maximum observed plasma concentration.
Part 1 and 2: Apparent Elimination Half-life (t1/2) of JNJ-70033093 | Up to 72 hours post dose
  Apparent elimination half-life associated with the terminal slope lambda(z) of the semilogarithmic drug concentration-time curve.

SECONDARY OUTCOMES:
Part 1 and 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2 Months
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.
Part 1 and 2: Number of Participants with Clinically Significant Changes in Vital Signs | Up to 2 Months
  Number of participants with clinically significant changes in vital signs including temperature (axillary), pulse rate, respiratory rate, blood pressure will be reported.
Part 1 and 2: Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to 2 Months
  Number of participants with abnormalities in ECG will be reported.
Part 1 and 2: Number of Participants with Clinically Significant Changes in Physical Examination | Up to 2 Months
  Number of participants with clinically significant changes in physical examination including height and body weight will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency